CLINICAL TRIAL: NCT05032313
Title: Evaluation of the Chronic Lymphoproliferative Diseases Limited Panel (BD OneFlow™ LST and OneFlow™ B-CLPD T1) on the BD FACSLyric™ Flow Cytometer Using Leftover, De-identified Specimens
Brief Title: Evaluation of the Chronic Lymphoproliferative Diseases Limited Panel on the BD FACSLyric™ Flow Cytometer
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CAS-OFLYRICLB-IVDR
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Lymphoproliferative Diseases (CLPD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Remnant/ Leftover specimens: Specimens that meet inclusion/exclusions criteria and are leftover from routine flow cytometry testing for hematological disorders.
  Interventions: Diagnostic Test: IUO CLPD Limited Panel

INTERVENTIONS:
Diagnostic Test: IUO CLPD Limited Panel — This Investigational Panel , comprised of 2 reagents , is intended for in vitro diagnostic use for qualitative flow-cytometric immunophenotyping of mature lymphocyte populations. These reagents are used as an aid in the differential diagnosis of hematologically abnormal patients having Chronic Lymphoproliferative Disease .

SUMMARY:
Multi-site, prospective performance study to determine equivalency between the investigational CLPD Limited Panel on the FACSLyric system versus the final clinical diagnosis.

DETAILED DESCRIPTION:
Hematology laboratories rely on flow cytometry technology (in addition to classic hematological methods) to aid in screening, diagnosing, and monitoring patients with hematological disorders. High speed and broad applicability of flow cytometry allows for the diagnosis. Currently, there are no consensus panels being used; consequently, the leukemia & lymphoma (L&L) testing remains a single-vial antibody being used with various in-house laboratory developed tests (LDTs) being used to test patient specimens. Furthermore, the analysis of flow cytometer generated data is not standardized and requires a high level of expertise and training for interpretation of complex data. Therefore, optimized and standardized immunostaining protocols for the diagnosis, classification, and prognostic sub-classification of hematological malignancies are needed.

This investigational reagent panel for chronic lymphoproliferative diseases (CLPD) is intended for in vitro diagnostic use for qualitative flow-cytometric immunophenotyping of mature lymphocyte populations on the BD FACSLyric flow cytometer . These reagents are used as an aid in the differential diagnosis of hematologically abnormal patients having, or suspected of having, B-cell CLPD, T-cell CLPD, and NK-cell CLPD.

Enrollment will occur at up to 8 investigational sites . Data will be acquired from Eligible remnant/leftover specimens on the BD FACSLyric flow cytometer and evaluated by site personnel and expert analysts .

The final diagnosis and the affected cell population will be determined by site standard of care .

Analysis of data will evaluate identification of normal vs abnormal cell population of the expert & site analysts as compared to the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Specimen collected/handled prior to enrollment in accordance with site policies and procedures.
2. Specimen with adequate volume (approximately 300 µL) to complete protocol tests.
3. Specimen is leftover PB, BM, or LN from routine flow cytometry laboratory testing for chronic lymphoproliferative disorders, other hematological disorders, non-hematological tumors (e.g., solid tumors), or other non-hematological disorders (non-malignant).
4. Specimen from newly diagnosed or relapsed subject.
5. Only one type of specimen, either PB, BM, or LN shall be enrolled per given subject.
6. Specimen is stored at room temperature, upon receipt by the site.
7. PB and BM specimens are collected in EDTA (K2 or K3) or heparin (sodium or lithium).
8. LN specimens collected in PBS, culture media (e.g., RPMI-1640), saline, or saline wrapped gauze at the discretion of the Investigator.
9. Age of specimen for PB and BM (time of collection to start of first pre-wash): ≤ 24 hours. (Note: No Age of specimen claim is being made for LN)
10. Specimens are from subjects irrespective of race, gender, and ethnicity.

Exclusion Criteria:

1. Specimen is from healthy subject.
2. Specimen is from subject undergoing any treatment for any form of L&L.
3. Specimen from subject <22 years of age.
4. Specimen is from subject with minimal residual disease (MRD) as determined by the site.
5. Specimen is from subject suspected of acute leukemia (e.g., T-ALL, BCP-ALL, AML) or myeloid dysplastic syndrome (MDS).
6. Visibly clotted specimen.
7. Visibly hemolyzed specimen.
8. Frozen specimen.
9. Refrigerated specimen.
10. Fixed specimen.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of evaluable 250 remnant/leftover peripheral blood, bone marrow, and lymph node specimens from routine flow cytometry laboratory testing for hematological disorders. Specimens from healthy subjects will be excluded.
  Specimens are from subjects irrespective of race, gender, and ethnicity. Specimen from subject >22 years of age .
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Comparison between expert analysts' determination of normal and abnormal specimen and final diagnosis | Age of specimen for PB and BM (time of collection to start of first pre-wash): ≤ 24 hours.
  Determine equivalence between the investigational OneFlow CLPD Limited Panel on FACSLyric system results analyzed by two independent experts versus the final clinical diagnosis for Normal (T-cell, B-cell, and NK-cell) or Abnormal (T-cell or B-cell or NK-cell) phenotype using leftover, hematologically abnormal specimens .
  Sensitivity and specificity are calculated

SECONDARY OUTCOMES:
Comparison between expert analysts' determination of normal and abnormal Peripheral Blood (PB) specimen and final diagnosis | Age of specimen for PB (time of collection to start of first pre-wash): ≤ 24 hours.
  Determine equivalence between the investigational OneFlow CLPD Limited Panel on FACSLyric system results analyzed by two independent experts versus the final clinical diagnosis for Normal or Abnormal phenotype using leftover, hematologically abnormal peripheral blood (PB) specimens.
  Sensitivity and specificity are calculated .

CONTACTS AND LOCATIONS:
Overall Officials: Imelda Omana-Zapata, MD, PHD, Study Director — Becton, Dickinson and Company
Locations (6):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Corepath Laboratories, San Antonio, Texas
- Champalimaud Foundation, Lisbon, Portugal
- University of Salamanca, Salamanca, Spain
- Kantonsspital Aarau, Aarau, Switzerland
- Cambridge university hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No